CLINICAL TRIAL: NCT01243385
Title: Metformin in Castration Resistant Prostate Cancer. A Multicenter Phase II Trial.
Brief Title: Metformin Hydrochloride as First-Line Therapy in Treating Patients With Locally Advanced or Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 08/09; SWS-SAKK-08/09; CDR0000688789 (Other: CDR0000688789)
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; hormone-resistant prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin (Other): Metformin at a target dose of 2 x 1000 mg daily Until progression, unacceptable toxicity or refusal
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin Lifelong follow-up at a target dose of 2 x 1000 mg daily Until progression, unacceptable toxicity or refusal
  Other Names: Metformin-Mepha

SUMMARY:
RATIONALE: Metformin hydrochloride may make some enzymes active. These enzymes may block other enzymes needed for cell growth and stop the growth of tumor cells.

PURPOSE: This phase II trial is studying the safety of giving metformin hydrochloride as first-line therapy in treating patients with locally advanced or metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the activity and safety of metformin hydrochloride as first-line therapy in patients with locally advanced or metastatic castration-resistant prostate cancer.

OUTLINE: This is a multicenter study.

Patients receive oral metformin hydrochloride twice daily on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Previously collected and post-treatment tumor tissue may be analyzed for PTEN status and PI3kinase-dependent pathway activation via immunohistochemistry. Blood samples may also be collected periodically and analyzed for biomarkers, pharmacogenetics, pharmacodynamics, pharmacokinetics.

After completion of study therapy, patients are followed up every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Locally advanced or metastatic disease with no curative therapy possible
* PSA progression defined as the following:

  * Increase in PSA of ≥ 25% (and an absolute increase of ≥ 2 ng/mL) over nadir value on hormonal therapy measured on 3 successive occasions at least 1 week apart

    * If the third measurement is not higher than the second, a fourth measurement will be taken and only if the fourth measurement is higher than the second, the patient may be enrolled
* PSA doubling time ≥ 55 days (if used to define progression, must not be older than 6 months)
* PSA < 114 ng/mL
* Testosterone level ≤ 1.7 nmol/L (≤ 50 ng/dL) after at least 1 hormonal treatment (orchiectomy or luteinizing hormone-releasing hormone [LHRH] agonist)
* Patients who have not undergone surgical castration must continue LHRH agonist therapy during study treatment
* Oligosymptomatic or asymptomatic in relation to disease
* No known or suspected CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Hemoglobin ≥ 90 g/L
* Neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* AST ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine clearance ≥ 60 mL/min
* Compliant and geographically proximal for proper staging and follow-up
* No previous malignancy within the past 2 years except for localized nonmelanoma skin cancer or Ta or Tis bladder cancer
* No history of diabetic ketoacidosis, diabetic coma, or pre-coma
* No known history of HIV, hepatitis B, or hepatitis C positivity
* No known hypersensitivity to the trial drug or any of its components
* No serious underlying medical condition that, in the judgment of the investigator, would impair the ability of the patient to participate in the trial (e.g., uncontrolled or acute severe infection, uncontrolled diabetes, advanced chronic obstructive pulmonary disease [COPD], or heart failure)
* No psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, or interfering with compliance for oral drug intake
* No known alcohol abuse

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 weeks since prior antiandrogen therapy and without withdrawal response
* At least 30 days since prior treatment in another clinical trial
* At least 4 weeks since prior major surgery
* At least 4 weeks since prior products known to affect PSA levels
* At least 2 weeks since prior local radiation
* No prior chemotherapy, radioisotopes, small molecules, or immunotherapy for prostate cancer
* No prior metformin hydrochloride
* No concurrent pharmacotherapy for diabetes mellitus
* No concurrent finasteride, dutasteride, ketoconazole, or abiraterone acetate
* No concurrent corticosteroids with an equivalent dose of > 7.5 mg of prednisolone
* No concurrent radiotherapy
* No bisphosphonates started after registration
* No concurrent drugs contraindicated for use with the trial drug according to the Swissmedic approved product information
* No other concurrent anticancer drugs
* No other concurrent experimental or investigational drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-12-23 (Actual); Primary Completion 2012-04-17 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at 12 weeks | at 12 weeks
  PFS is defined as the absence of disease progression or death at 12 weeks after start of treatment.

SECONDARY OUTCOMES:
PFS at 24 weeks | at 24 weeks
  PFS is defined as the absence of any disease progression or death at 24 weeks after start of treatment
Clinical benefit rate | at 12 weeks and 24 weeks
  Clinical benefit is defined as SD by imaging and symptoms - with or without PSA progression
Adverse events | from start of treatment until progression or death of any cause
  All AEs will be assessed according to NCI CTCAE v4.0
Prostate-specific antigen (PSA) response | (50% and 30%, best and at 12 weeks)
  50 % PSA response is defined as a decrease in PSA level of at least 50 % (compared to baseline PSA).
  30 % PSA response is defined as a decrease in PSA level of at least 30 % (compared to baseline PSA).
  Best response is defined as the percentage of change in PSA from baseline to the maximum decline in PSA at any point under treatment at 12 weeks or later. If there is a steady increase after baseline, the best response is defined as the percentage of change in PSA from baseline to the minimum increase in PSA at any point under treatment at 12 weeks or later.
Changes in PSA doubling time | after 12 weeks, after 24 weeks and at best PSA response
  PSA-DT is calculated from the natural log of 2 divided by the slope of the relationship between the log of PSA and the time of PSA measurement for each patient.
Tumor response of measurable disease according to RECIST v 1.1 criteria | after 12 weeks of treatment
  For patients with measurable disease at baseline RECIST v1.1 will be used to define CR, PR, SD and PD.
Tumor assessment of bone lesions | at 12 weeks
  Bone metastases can be assessed by radionuclide bone scan.
Overall survival | from registration until death
  OS will be calculated from registration until death

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rothermundt, MD, Study Chair — Cantonal Hospital of St. Gallen; Richard Cathomas, MD, Study Chair — Kantonsspital Graubuenden; Silke Gillessen, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (9):
- Switzerland (9):
  - Kantonsspital Aarau, Aarau
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital Luzern, Luzerne
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rothermundt C, Hayoz S, Templeton AJ, Winterhalder R, Strebel RT, Bartschi D, Pollak M, Lui L, Endt K, Schiess R, Ruschoff JH, Cathomas R, Gillessen S. Metformin in chemotherapy-naive castration-resistant prostate cancer: a multicenter phase 2 trial (SAKK 08/09). Eur Urol. 2014 Sep;66(3):468-74. doi: 10.1016/j.eururo.2013.12.057. Epub 2014 Jan 4. PMID 24412228